CLINICAL TRIAL: NCT05695287
Title: The Effects of Sevoflurane, Isoflurane and Propofol on the Hemodynamic, Body Energy Expenditure During Cardiac Surgery in Adults: a Randomized Clinical Trial
Brief Title: The Effects of Sevoflurane, Isoflurane and Propofol During Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Bekzat Baiterek, Clinical Professor, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease; Mitral Valve Insufficiency; Aortic Valve Insufficiency
Keywords: heart valve; CHD; sevoflurane; propofol; isoflurane
MeSH Terms: conditions — Coronary Artery Disease; Mitral Valve Insufficiency; Aortic Valve Insufficiency | interventions — Propofol; Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Other): Anesthesia
  Interventions: Drug: Propofol
- Isofluran (Other): Anesthesia
  Interventions: Drug: Isoflurane
- Sevofluran (Other): Anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 4-6 mg/kg/h intravenously on a perfusor
  Other Names: Propofol;
  Arms: Propofol
Drug: Isoflurane — Isoflurane
  Other Names: В качестве анестетика использовали изофлуран - 1,1-1,2 ПДК.
  Arms: Isofluran
Drug: Sevoflurane — Sevoflurane
  Other Names: в качестве анестетика использовали севофлуран в дозе - 1,7-1,9 ПДК.
  Arms: Sevofluran

SUMMARY:
Abstract Anaesthetic support for cardiac surgery significantly influences the course of the intraoperative period and the success of the postoperative period. Total intravenous anaesthesia and inhalation anaesthesia are the traditional methods of anaesthesia in cardiac surgery. However, there are few studies assessing the effectiveness of surgical aggression protection in cardiac surgery.

Objectives: To study the effectiveness of body protection against surgical aggression by TIVA and inhalational anaesthesia in cardiac surgery.

Materials and methods. The examination and treatment data of 89 patients were included in the study. All patients underwent coronary artery bypass grafting, mitral valve replacement/plasty, aortic valve replacement cardiopulmonary bypass conditions.

The patients were divided into 2 groups according to the type of disease: the first (1) group with coronary heart disease. The second (2) group with valvular heart disease. There were 65 patients in the first group and 22 in the second. Both groups were divided into 3 subgroups according to the type of anaesthesia: patients anaesthetised with propofol, with sevoflurane, with isoflurane.

DETAILED DESCRIPTION:
All patients were divided into 2 groups according to the type of disease: the first (1) group with coronary heart disease. The second (2) group with valvular heart disease. There were 65 patients in the first group and 22 in the second. Both groups were divided into 3 subgroups according to the type of anaesthesia: patients anaesthetised with propofol, with sevoflurane, with isoflurane.

The study was conducted in 5 stages:

1. Initial haemodynamic parameters and oxygen transport function of the patient's blood before anaesthesia were determined;
2. after tracheal intubation;
3. Before the CPB;
4. after the CPB;
5. The post-operative period until the patient is extubated. Before induction into anaesthesia, haemodynamic monitoring was started on admission to the operating theatre using a Nihon Kohden monitor (Japan). The right radial artery was catheterised for invasive monitoring of systemic arterial pressure and arterial blood sampling, and a catheter was then inserted into the central jugular vein (under ultrasound machine control) and guided into the right atrium for mixed venous blood sampling.

Cardiac stroke volume was determined by transthoracic echocardiography (CS=end diastolic volume - end systolic volume). Cardiac output (CO=CS x heart rate), cardiac index (CI=CO/body surface area) were determined. We determined blood oxygen content using the formula CaO2 (arterial ABB) and CvO2 (central mixed venous ABB) = [(1.34 × Hb × SO2) + (PO2 × 0.031)] / 100. Arteriovenous difference = CaO2-CvO2. Oxygen delivery was determined using the formula (DO2 = CI* CaO2). Oxygen consumption (VO2 = Cardiac index (CI)*AVD or VO2 = CO × (CaO2 - CvO2) ~ CO × Hb × 1.34 × (SaO2 - SvO2) / 100).

In the second stage, after tracheal intubation, indirect calorimetry was used to determine VO2, energy expenditure during anaesthesia using a Spirometry device (Oxford, UK), which was connected to an endotracheal tube and continuously showed oxygen demand and energy expenditure. A transesophageal echocardiography sensor was used to determine cardiac output. Additionally, the cardiac output was determined by Fick's formula in patients with CHD. The same tests (cardiac output, cardiac index, consumption, oxygen delivery, energy expenditure) were performed in the third and fourth stages of anaesthesia. In the last stage, the consumption of muscle relaxants and opioid analgesics was calculated to assess the pharmaco-efficiency of anaesthetics. The time of extubation and the time of transfer of the patient to the specialist department were determined.

All patients continued antihypertensive medication both before and on the day of surgery to prevent the development of withdrawal syndrome and to reduce the risk of perioperative myocardial ischaemia.

All patients in both groups were anesthetized with fentanyl at a dose of 5-7 µg/kg, ketamine 1.5-2 mg/kg, and propofol 1-1.5 mg/kg intravenously fractionally. Pipecuronium bromide 0.04-0.07 mg/kg was used as muscle relaxant in all patients. To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 4-6 mg/kg/h intravenously on a perfusor (BBRAUN). In Group 2, sevoflurane was used as an anaesthetic in a dose of - 1.7-1.9 MAC. In Group 3 isoflurane was used as the anesthetic in the dose of 1.1-1.2 MAC. Fentanyl 100 µg intravenously was administered fractionally in all groups to increase heart rate and blood pressure, and pipecuronium bromide 2 mg intravenously for myorelaxation. During CPB, propofol at a dose of 6 mg/kg/h intravenously via perfusion was used in all patients in all groups. Anaesthesia regimen: fentanyl 100 µg IV every 30 min; myorelaxant pipecuronium bromide 2 mg every 40-60 min. Norepinephrine solution was administered at a dose of 0.07 µg/kg/min intravenously on perfusion and dobutamine 5 µg/kg/min after CPB in all patients at the same dosages in all groups.

ELIGIBILITY:
Inclusion Criteria:

* • The age is between 40-60 years old;

  * Mitral valve insufficiency grade 3-4;
  * Aortic valve insufficiency grade 3-4;
  * Participants of both sexes will be included in the study;
  * Signed informed consent.

Exclusion Criteria:

* • pregnancy (risk to the baby and the mother)

  * allergenic patients (anaphylactic shock).
  * vulnerable groups.
  * current congestive heart failure;
  * current unstable angina pectoris;
  * preoperative hemodynamic instability, defined as the use of vasopressors;

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
cardiac index | 1 year
  cardiac index (CI=CO/body surface area
Oxygen consumption | 1 year
  oxygen consumption (VO2 = Cardiac index *AVD or VO2 = CO × (CaO2 - CvO2) ~ CB × Hb × 1,34 × (SaO2 - SvO2) / 100)
Oxygen delivery | 1 year
  The oxygen delivery was found by formula (DO2 = CI* CaO2)
cardiac stroke | 1 year
  The cardiac stroke (CS) volume was determined by transthoracic echocardiography (CS =end diastolic volume-end systolic volume).

CONTACTS AND LOCATIONS:
Overall Officials: Alibek Kh Mustafin, Professor, Study Director — Astana Medical University
Locations (1):
- Bekzat, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No